CLINICAL TRIAL: NCT07067944
Title: The Preventive Role of Prophylactic Perioperative Infusion of Ephedrine Versus Noradrenaline in Patients Undergoing Cesarean Delivery Under Spinal Anesthesia: A Randomized, Prospective Double-blinded Study
Brief Title: Prophylactic Perioperative Infusion of Ephedrine Versus Noradrenaline in Patients Undergoing Cesarean Delivery Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hadeer Gamal Fouda, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264MS146/4/23
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Perioperative Infusion; Ephedrine; Noradrenaline; Cesarean Delivery; Spinal Anesthesia
MeSH Terms: interventions — Ephedrine; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The parturient will receive ephedrine infusion immediately before intrathecal injection till delivery of the baby at a dose of 4mg /min.
  Interventions: Drug: Ephedrine
- Group B (Experimental): The parturient will receive noradrenaline infusion immediately before intrathecal injection till delivery of the baby at a dose of 4 microgram/minute.
  Interventions: Drug: Noradrenaline

INTERVENTIONS:
Drug: Ephedrine — The parturient will receive ephedrine infusion immediately before intrathecal injection till delivery of the baby at a dose of 4mg /min.
  Arms: Group A
Drug: Noradrenaline — The parturient will receive noradrenaline infusion immediately before intrathecal injection till delivery of the baby at a dose of 4 microgram/minute.
  Arms: Group B

SUMMARY:
This study aimed to compare the effects of prophylactic ephedrine and nor-epinephrine infusion on maternal hemodynamics and neonatal outcomes following spinal anesthesia in cesarean deliveries.

DETAILED DESCRIPTION:
Neuraxial anesthesia for cesarean delivery (CD) has significantly reduced maternal mortality by avoiding Manipulation of the airway, the mother being awake, and promoting early bonding of mother and child, adequate Postoperative analgesia, and quicker maternal recovery.

Systemic vascular resistance decreases as a result of a reduction in sympathetic tone of the arterial circulation, leading to peripheral arterial vasodilation, the extent of which depends on the number of spinal segments involved. Other theories are proposed to explain hypotension during spinal anesthesia, among them: 1)direct depressive circulatory effect of local anesthetics, 2) relative adrenal insufficiency, 3) skeletal muscle paralysis, 4) ascending medullary vasomotor block, and 5) concurrent mechanical respiratory insufficiency. Loss of sympathetic input to the heart, leaving vagal parasympathetic innervations unopposed, and a decrease in cardiac preload are the main reasons for bradycardia during spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 21 years.
* American Society of Anesthesiologists Physical Status II and III.
* Full-term singleton pregnant women scheduled for elective cesarean section under spinal anesthesia.

Exclusion Criteria:

* Morbid obesity [body mass index (BMI)>40].
* Diabetes Mellitus.
* Severe cardiovascular disease.
* Hypertensive disorders of pregnancy.
* Chronic kidney disease.
* Non-assuring fetal status.
* Peripartum bleeding.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing cesarean delivery
Enrollment: 100 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Maternal systolic blood pressure | 10 minutes after induction of spinal anesthesia
  Maternal systolic blood pressure was recorded 10 minutes after induction of spinal anesthesia.

SECONDARY OUTCOMES:
Heart rate | Intraoperatively
  Intraoperative heart rate was recorded after spinal anesthesia induction.
Number of needed rescue boluses of vasopressors | After induction of spinal anesthesia (Up to 2 hours)
  Number of needed rescue boluses of vasopressors to keep hemodynamic stability after spinal anesthesia induction.
Incidence of adverse events | 2 hours after induction of spinal anesthesia
  Incidence of adverse events such as nausea and vomiting were recorded.
APGAR score | 5 minutes after delivery
  APGAR score was recorded at 1 and 5 minutes after delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.